CLINICAL TRIAL: NCT06818370
Title: The Effect of Coconut Oil on Alopecia in Women Receiving Doxorubucin-Cycylophosphamide Treatment for Breast Cancer
Brief Title: The Effect of Coconut Oil on Alopecia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, İsmail DAKDEVİR, Nurse, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ankara Onkoloji EAH
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Alopecia; Breast Cancer; Coconut Oil
MeSH Terms: conditions — Breast Neoplasms; Alopecia | interventions — Coconut Oil

STUDY DESIGN:
Intervention Model Description: It will be conducted in a randomized controlled experimental design.
Who Masked: Participant
Masking Description: Patients with breast cancer in the experimental and control groups will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): At the beginning of the study,patients will be asked to fill out an individual information form containing demographic information and disease process before the first chemotherapy application.The coconut oil application protocol will be explained to the patients in the experimental group and 10 milliliters of coconut oil will be applied to the hair follicles once a week. Alopecia assessment will be done every week.
  Interventions: Other: Coconut Oil
- Control Group (No Intervention): At the beginning of the study,patients will be asked to fill out an individual information form containing demographic information and disease process before the first chemotherapy application. Patients in the control group will be asked not to apply anything to their hair. In each subsequent week, the presence of hair loss of the patients will be evaluated with the alopecia evaluation scale.

INTERVENTIONS:
Other: Coconut Oil — The coconut oil application protocol will be explained to the patients in the experimental group and 10 milliliters of coconut oil will be applied to the hair follicles once a week. Alopecia assessment will be done every week.
  Arms: Experimental group

SUMMARY:
İn this study will be conducted to evaluate the effect of coconut oil on alopecia in 86 female breast cancer patients treated at Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital between 01.02.2025-31.12.2025.

DETAILED DESCRIPTION:
Cancer is a disease in which the cells in our body multiply uncontrollably and develop by metastasizing, and the symptoms, course and consequences of the disease can show complex qualities in each patient. Cancer treatments have benefits and harms. One of these side effects is alopecia.

Alopecia due to cancer treatments is a condition of hair loss, partial or complete, usually temporary but rarely permanent.

In chemotherapy-induced alopecia, the hair follicle is damaged due to the pause in the anagen phase and causes the hair to break off spontaneously during activities such as washing and brushing the hair.

Various scales are used in the evaluation of alopecia due to cancer treatments, such as the National Cancer Institute Common Terminology Criteria for Side Effects and the Dean Alopecia Scale.

Some applications are made to prevent and treat alopecia. These include strategies and pharmacological applications to physically reduce the amount of medication given to the hair follicle.

Coconut oil helps regrow damaged hair. It provides essential proteins necessary for hair and softens the scalp and hair.

In the literature, it has been observed that studies showing the effects of coconut oil for the prevention and treatment of alopecia are insufficient. This study will be conducted on 86 breast cancer patients to determine the effect of coconut oil on the development of alopecia.

ELIGIBILITY:
Inclusion Criteria:

* • To have been diagnosed with breast cancer.

  * The chemotherapy treatment plan should be planned as the Doxorubicin-Cyclophosphamide protocol.
  * Volunteer to participate in the study.
  * Be 18 years of age or older.
  * Being a woman.

Exclusion Criteria:

* • Having any health problem or disability that prevents communication (vision-hearing problems, neurological, psychiatric diseases).

  * Planning other treatments other than the Doxorubicin-Cyclophosphamide protocol for the treatment of breast cancer.
  * Not volunteering to participate in the study.
  * Having previously experienced any disease/skin problem that causes hair loss.
  * Having received chemotherapy before.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 86 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
National Cancer Instute (NCI) Common Terminology Criteria for Adverse Events (CTCAE); Alopecia | 1-12 WEEK
  Grade 1; Hair loss of <50% of normal for that individual that is not obvious from a distance but only on close inspection; a different hair style may be required to cover the hair loss but it does not require a wig or hair piece to camouflage Grade 2; Hair loss of >=50% normal for that individual that is readily apparent to others; a wig or hair piece is necessary if the patient desires to completely camouflage the hair loss; associated with psychosocial impact

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Onkoloji Eğitim ve Araştırma Hastanesi, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No